CLINICAL TRIAL: NCT05736601
Title: Early Outcomes of MAKO Medial Unicompartmental Knee Arthroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Other Study IDs: 202203201
Record Dates: First submitted 2023-01-31; First posted 2023-02-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- UKA MAKO: Prospective group- Patient Reported Outcomes (PROs) will be assessed using the FocusMotion app survey
  Interventions: Device: focus motion knee brace
- TKA MAKO: Control group-Already collected data on patient reported out comes using the FocusMotion app survey
  Interventions: Device: focus motion knee brace

INTERVENTIONS:
Device: focus motion knee brace — knee brace that captures knee motion

SUMMARY:
To determine if robotically-assisted UKA results in more consistent and improved component positioning and better patient reported outcome scores compared to manual TKA and MAKO TKA.

DETAILED DESCRIPTION:
The purpose of this study is to determine the early clinical and radiographic outcomes of robotically-assisted medial unicompartmental knee arthroplasty (mUKA) with the MAKO surgical robot using the Restoris MCK Partial Implant System. The primary end point will be the mean weekly VAS pain score during the first four weeks postoperatively. The results of this study may be compared to those of previously studied cohorts of patients from this institution who underwent manual total knee arthroplasty (TKA) with the Triathlon Knee System as well as robotically-assisted total knee arthroplasty with the MAKO surgical robot using the Triathlon Knee System

ELIGIBILITY:
Inclusion Criteria:

A. Unilateral primary medial unicompartmental knee arthroplasty

B. Age 18 years of age or older

C. Willing to sign informed consent

D. Willing to return for all follow-up visits

E. Smartphone or tablet device capable of running the FocusMotion platform

Exclusion Criteria:

A. BMI > 40

B. Personal history of DVT or PE

C. Inflammatory arthritis

D. Peripheral vascular disease

E. Opioid use greater than 5 days per week

F. Nonsteroidal anti-inflammatory allergy

G. Walking aid for musculoskeletal or neurologic issue other than operative joint

H. Bilateral medial unicompartmental knee arthroplasty

I. Patient with an active infection or suspected infection in the operative joint

J. The absolute and relative contraindications stated in the FDA cleared labeling for the device

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants 18 years and older who have chosen to partial knee surgery using the mako robotic system.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient reported Questionnaires for weekly VAS pain scores up weekly | 1 year
  Patients will assess their weekly pain scores by filling out patient reported outcomes.

SECONDARY OUTCOMES:
Patient will track their Opioid Consumption use by filling out a chart weekly | 3 months
  Patients will report their weekly use by Opioid Consumption filling out a patient diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University Medical School, St Louis, Missouri, United States

REFERENCES:
- [Background] Kayani B, Konan S, Tahmassebi J, Pietrzak JRT, Haddad FS. Robotic-arm assisted total knee arthroplasty is associated with improved early functional recovery and reduced time to hospital discharge compared with conventional jig-based total knee arthroplasty: a prospective cohort study. Bone Joint J. 2018 Jul;100-B(7):930-937. doi: 10.1302/0301-620X.100B7.BJJ-2017-1449.R1. PMID 29954217
- [Result] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Result] Kazarian GS, Barrack TN, Okafor L, Barrack RL, Nunley RM, Lawrie CM. High Prevalence of Radiographic Outliers and Revisions with Unicompartmental Knee Arthroplasty. J Bone Joint Surg Am. 2020 Jul 1;102(13):1151-1159. doi: 10.2106/JBJS.19.01277. PMID 32618922
- [Result] Nam D, Berend ME, Nunley RM, Della Valle CJ, Berend KR, Lombardi AV, Barrack RL. Residual Symptoms and Function After Unicompartmental and Total Knee Arthroplasty: Comparable to Normative Controls? J Arthroplasty. 2016 Oct;31(10):2161-6. doi: 10.1016/j.arth.2016.02.064. Epub 2016 Mar 10. PMID 27067170
- [Result] Lee BS, Cho HI, Bin SI, Kim JM, Jo BK. Femoral Component Varus Malposition is Associated with Tibial Aseptic Loosening After TKA. Clin Orthop Relat Res. 2018 Feb;476(2):400-407. doi: 10.1007/s11999.0000000000000012. PMID 29389790